CLINICAL TRIAL: NCT01518868
Title: A Study to Evaluate the Feasibility of a High Add Multi Focal Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 743E
Record Dates: First submitted 2012-01-24; First posted 2012-01-26 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational contact lens (Experimental): multifocal high add soft contact lens
  Interventions: Device: Investigational contact lens
- PureVision contact lens (Active Comparator): Multi-focal contact lens
  Interventions: Device: PureVision contact lens

INTERVENTIONS:
Device: Investigational contact lens — Worn on a daily wear basis for one week.
  Arms: Investigational contact lens
Device: PureVision contact lens — Worn on a daily wear basis for one week
  Arms: PureVision contact lens

SUMMARY:
The objective of this study is to evaluate the product performance of the investigational multifocal high add soft contact lens compared with PureVision Multi-focal contact lens on a daily wear basis.

ELIGIBILITY:
Inclusion Criteria:

* Have physiologically normal anterior segments
* Be adapted wearers of soft contact lenses and wear a lens in each eye.
* Be presbyopic and require near add correction in each eye.
* Be an adapted monovision or multifocal contact lens wearer or be an adapted spherical lens wearer who also uses spectacles for near vision correction.
* Have no active ocular disease or allergic conjunctivitis.
* Must not be using any topical ocular medications.
* Must habitually use a lens care product for lens cleaning, disinfecting, and storage.

Exclusion Criteria:

* Any Grade 2 or greater finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Anisometropia (spherical equivalent) of greater than 2.00 D.
* Any systemic disease affecting ocular health.
* Using any systemic or topical medications that will affect ocular physiology or lens performance.
* Allergic to any component in the study products.
* Ocular astigmatism of greater than 1.00 D in either eye.
* Have had any corneal surgery (ie, refractive surgery).
* Uses AMO Ultra Care as their habitual lens care regimen.
* Is a toric contact lens wearer.
* Have worn gas permeable (GP) contact lenses within last 30 days or PMMA lenses within last 3 months.
* An active ocular disease (for example but not limited to papillary conjunctivitis, any conjunctivitis: viral, bacterial, allergic), any corneal infiltrative response or are using any ocular medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly J Barna, CCRA, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 126 participants (252 eyes) were enrolled. One-half of the participants were randomized to receive the investigational contact lens during the first crossover period, and the other half were randomized to receive the PureVision contact lens during the first crossover period. The participants crossed over to the other group at 1 week.
Groups:
- Investigational Contact Lens Then PureVision Contact Lens: multifocal high add soft contact lens
  Investigational contact lens: Worn on a daily wear basis for one week.
  Multi-focal contact lens PureVision contact lens: Worn on a daily wear basis for one week
- PureVision Contact Lens: Multi-focal contact lens then Investigational Contact Lens
  PureVision contact lens: Worn on a daily wear basis for one week
  multifocal high add soft contact lens Investigational contact lens: Worn on a daily wear basis for one week.
Period: Overall Study
Arm/Group | Investigational Contact Lens Then PureVision Contact Lens | PureVision Contact Lens
Started | 63 | 63
Completed | 59 | 59
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: Demography was collected for 124 eligible, dispensed participants. Participants received both treatment groups in this cross-over study.
Groups:
- Overall: Participants received both treatment groups in this cross-over study.
Arm/Group | Overall
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Visual acuity was assessed by distance high contrast logarithm of the minimum angle of resolution (logMAR).
Time Frame: At 2 weeks follow up
Population: There were 238 eyes assessed for visual acuity for this outcome measure. Participants/eyes received both treatment groups.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eye
Arm/Group | Investigational Contact Lens | PureVision Contact Lens
Number analyzed (Participants) | 119 | 119
Number analyzed (eye) | 238 | 238
logMAR | 0.079 (0.102) | 0.090 (0.091)

2. Secondary Outcome: Symptoms/Complaints
Description: Symptoms/complaints were assessed on a scale from 0 to 100, with 0 denoting unfavorable symptoms/complaints.
Time Frame: At 2 weeks follow up
Population: There were 238 eyes assessed for symptoms/complaints for this outcome measure. Participants/eyes received both treatment groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Investigational Contact Lens | PureVision Contact Lens
Number analyzed (Participants) | 119 | 119
Number analyzed (eyes) | 238 | 238
score on a scale
  Burning/stinging upon insertion | 95.6 (8.9) | 92.5 (14.7)
  Comfort upon insertion | 89.4 (17.0) | 81.5 (25.0)
  Comfort at end of day | 75.3 (25.4) | 64.9 (28.8)
  Overall comfort | 81.6 (20.3) | 70.5 (26.7)
  Dryness | 80.3 (20.3) | 73.3 (26.4)
  Itchiness | 91.9 (13.8) | 86.8 (22.1)
  Redness | 91.4 (14.4) | 86.9 (23.0)
  Distance vision | 67.7 (29.8) | 59.3 (30.8)
  Vision at intermediate distance | 80.5 (22.5) | 70.3 (25.8)
  Vision at near distance | 65.0 (30.0) | 58.8 (30.8)
  Overall vision | 66.7 (25.4) | 56.2 (27.5)
  Ease of handling/insertion | 86.5 (20.4) | 84.3 (21.7)
  Ease of handling/removal | 88.6 (16.3) | 86.2 (19.6)
  Overall impression | 73.3 (23.5) | 61.1 (29.9)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse events (AEs) were not coded. Therefore, source vocabulary is not applicable. A total of 126 participants (262 eyes) were assessed for AEs. Participants/eyes received both treatment groups in this cross-over study.
Groups:
- Investigational Contact Lens: multifocal high add soft contact lens
  Investigational contact lens: Worn on a daily wear basis by adapted monovision soft contact lens wearers for one week.
  Investigational contact lens: Worn on a daily wear basis by adapted multifocal soft contact wearers for one week.
  Investigational contact lens: Worn on a daily wear basis by adapted spherical soft contact lens wearers who may also use spectacles for near vision correction for one week
- PureVision Contact Lens: Multi-focal contact lens
  PureVision contact lens: Worn on a daily wear basis by adapted monovision soft contact lens wearers for one week
  PureVision contact lens: Worn on a daily wear basis by adapted multifocal soft contact wearers for one week.
  PureVision contact lens: Worn on a daily wear basis by adapted spherical soft contact lens wearers who may also use spectacles for near vision correction for one week
Arm/Group | Investigational Contact Lens | PureVision Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/126
Other Adverse Events (participants affected / at risk) | 0/126 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.